CLINICAL TRIAL: NCT00546221
Title: Pragmatic Randomised Controlled Trial of a Preferred Intensity Exercise Programme to Improve Physiological and Associated Psychological, Social, and Wellbeing Outcomes of Women Living With Depression
Brief Title: Promoting Wellbeing for Women With Depression: A Pragmatic Randomised Controlled Trial (RCT) of an Exercise Programme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Burdett Trust for Nursing (Other); Nottinghamshire Healthcare NHS Trust (Other Government); Nottingham City Primary Care Trust (Unknown); Nottinghamshire County Teaching Primary Care Trust (Unknown)
Responsible Party: Mr Paul Cartledge, University of Nottingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07105; Funder's ID: 293/350; Ethics ref ID: 07/H0401/110
Record Dates: First submitted 2007-10-17; First posted 2007-10-18 (Estimated); Last update posted 2011-03-03 (Estimated); Status verified 2011-03

CONDITIONS: Depression
Keywords: Depression; Mental health; Exercise; Prescribed exercise; Physical health; Social wellbeing
MeSH Terms: conditions — Depression; Psychological Well-Being; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psychosocial support (Experimental): Comprising 22 participants engaging in the experimental exercise programme, exercising with psychosocial support.
  Interventions: Behavioral: Psychosocial support exercise programme
- Prescribed exercise (Active Comparator): Comprising 21 participants engaging in a programme of typical prescribed exercise.
  Interventions: Behavioral: Prescribed exercise

INTERVENTIONS:
Behavioral: Psychosocial support exercise programme — The experimental arm will experience 12 sessions of intervention, at a rate of three sessions a week for four weeks, exercising in groups of ten women. Each session will comprise: fifteen minutes of psychosocial and motivational support, run by a qualified rehabilitation psychologist and overseen by a qualified health psychologist; a half hour preferred intensity exercise session run by a qualified sports physiotherapist. Participants preferred intensity (chosen exertion level) will be established using the Borg RPE scale (Borg G 1998).
  Arms: Psychosocial support
Behavioral: Prescribed exercise — This group will experience 12 sessions of intervention, at a rate of three sessions a week for four weeks, exercising in groups of ten women. Each session will be an half hour exercise session, at a typically (GP) prescribed level, designed in accordance with national guidelines and run by a qualified sports physiotherapist.
  Arms: Prescribed exercise

SUMMARY:
The investigators want to find out if their specially designed exercise programme will be more successful at helping women with depression to feel better than a basic programme will, by measuring the effect the programme has on mood, physical health, and social wellbeing. Their specially designed exercise programme will involve physical exertion at the participants' chosen level of intensity (how hard the body has to work during exercise), and will include motivational support. By contrast, the basic exercise programme will be at an intensity recommended by national guidelines, of the type that may be prescribed by a general practitioner (GP), and will include no extra motivational support.

ELIGIBILITY:
Inclusion Criteria:

* Living with depression
* Aged 18 (age at first session of programme)
* Female
* Living in the community
* Resident within Nottinghamshire (personal address has Nottinghamshire postcode)

Exclusion Criteria:

* Women who, at the time of the study, are unable to participate on account of any injury or physical health problem that precludes their participation
* Women participating in research that may undermine the scientific basis of the study

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2007-11; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is score on the BDI-II (Beck Depression Inventory version 2). | At the plenary session of the programmes.

SECONDARY OUTCOMES:
Resting heart rate. | At the plenary session of the programmes.
GHQ12. | At the plenary session of the programmes.
The SF-12vII. | At the plenary session of the programmes.
The Rosenberg self-esteem scale. | At the plenary session of the programmes.
Quality of life in depression scale. | At the plenary session of the programmes.
The multidimensional scale of perceived social support. | At the plenary session of the programmes.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Callaghan, RN BSc MSc PhD CPsychol, Principal Investigator — University of Nottingham; Elizabeth B Khalil, BSc MSc PhD (Cant.), Principal Investigator — University of Nottingham
Locations (3):
- United Kingdom (3):
  - Nottingham City Primary Care Trust, Nottingham, Nottinghamshire
  - Nottinghamshire County Teaching Primary Care Trust, Nottingham, Nottinghamshire
  - Nottinghamshire Healthcare NHS Trust, Nottingham, Nottinghamshire

REFERENCES:
- [Derived] Callaghan P, Khalil E, Morres I, Carter T. Pragmatic randomised controlled trial of preferred intensity exercise in women living with depression. BMC Public Health. 2011 Jun 12;11:465. doi: 10.1186/1471-2458-11-465. PMID 21663696
- See also: University of Nottingham, School of Nursing Mental Health Research Group — http://www.nottingham.ac.uk/nmp/research/mental-health/index.php
- See also: project website — http://www.nottingham.ac.uk/nursing/exercise_wellbeing/index.php